CLINICAL TRIAL: NCT04911088
Title: Does Calibration of Electromyography Guided by State Entropy Improve Measurement Precision
Brief Title: Electromyographic Calibration Guided by Depth of Anesthesia
Acronym: CELESTE
Status: Completed | Type: Observational
Sponsor: University Hospital Ulm (Other)
Collaborators: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Manfred Blobner, Professor of Anesthesiology, University Hospital Ulm
Other Study IDs: CELESTE-01
Record Dates: First submitted 2021-05-27; First posted 2021-06-02 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Neuromuscular Blockade
Keywords: electromyography; calibration; residual paralysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Analgesic calibration: Participants will receive calibration of electromyography at state entropy of 90.
- Sedated calibration: Calibration will be started at state entropy of 70.
- No calibration: Participants will not receive calibration of electromyography. Measurements will start simultaneously to the standard electromyography with a default current of 60mA at state entropy of 50.

SUMMARY:
The goal of the CELESTE study is to evaluate whether calibration of EMG is needed for reliable interpretation of neuromuscular function and if so, to identify the minimal necessary depth of anesthesia.

DETAILED DESCRIPTION:
Neuromuscular monitoring is used to document neuromuscular function intra-operatively. Failure to restore neuromuscular function prior to extubation results in residual neuromuscular blockade which is associated with increased postoperative morbidity and mortality. It is essential to document baseline neuromuscular function before administration of the neuromuscular blocking agent. However, during anesthesia induction, neuromuscular monitoring is rarely calibrated due to its time-consuming nature coinciding with the patients' loss of consciousness.

The CELESTE trial is a randomized, prospective, observational proof-of-concept study. We plan to enroll sixty adult participants scheduled for elective non-cardiac surgery requiring general anesthesia with moderate neuromuscular blockade. Participants will be randomized into three electromyography (EMG) calibration groups: based on state entropy ("depth of anesthesia"), group 1 will receive "analgesic calibration", group 2 "sedated calibration", and group 3 "no calibration". Participants will be randomly allocated to receive calibration at a certain depth of anesthesia. All participants will receive a standard EMG performed on the contralateral arm. Standard EMG will be calibrated at state entropy of 50.

ELIGIBILITY:
Inclusion Criteria:

* signed informed written consent
* BMI 17.5-30 kg/m^2
* ASA <= 3
* supine positioning during surgery with intraoperative access to both arms
* absence of allergy to muscle relaxants and reversal agents
* absence of neuromuscular disease

Exclusion Criteria:

* ambulatory patients for whom discharge is planned within 12 hours of anaesthesia
* patients undergoing minor surgical
* procedures scheduled outside the operating room
* patients who are endotracheally intubated prior to surgery
* pregnancy
* indication for rapid sequence induction
* patients undergoing arm surgery
* patients with preceding injuries impairing muscle or nerve function of the arm (e.g., finger amputation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The CELESTE study will be performed in adult patients scheduled for elective non-cardiac surgery requiring general anesthesia and moderate neuromuscular blockade.
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2022-01-16 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Precision of TOF measurements | intraoperative
  repeatability coefficient

SECONDARY OUTCOMES:
Tolerance interval of TOF ratios | intraoperative
Agreement of EMG calibration group TOF and standard TOF | intraoperative
  Agreement of both calibration group EMG and standard EMG regarding the decision whether complete neuromuscular recovery is given based on a TOF ratio of >0.9 or >0.95, respectively.
Time difference between calibration group TOF and standard TOF to complete recovery | intraoperative
  Time difference between calibration group EMG and the standard EMG reaching a TOF ratio >0.9 or >0.95, respectively.
Recall of calibration | postoperative day 1
Discomfort with calibration | postoperative day 1

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Blobner, MD PhD, Principal Investigator — Department of Anesthesiology and Intensive Care Medicine, University of Ulm, Ulm, Germany.
Locations (1):
- University Hospital Ulm, Ulm, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Scheffenbichler FT, Ulm B, Borgstedt L, Scholze A, Kretsch N, Zia N, Friedrich V, Marb M, Schaller SJ, Jungwirth B, Blobner M. Precision of electromyography according to the calibration approach of neuromuscular monitoring: a randomised prospective agreement study. J Clin Monit Comput. 2025 Oct;39(5):1047-1056. doi: 10.1007/s10877-025-01304-z. Epub 2025 May 28. PMID 40437152